A Pilot Trial Comparing NicoBloc to Nicotine Lozenges: Initial Acceptability and Feasibility Trial 2/2/2022 NTC:300001370

## **Data Analytic Approach**

Participant screening, baseline eligibility, baseline attendance, study eligibility, and retention rates throughout the study were calculated overall and per time point. Retention rates between groups at each time point and other dichotomized variables such as adherence were assessed using Chi-Square analyses. Participant demographics and baseline smoking characteristics were assessed, and group differences examined using measures of effect size (Cramer's *V* and Cohen's *d*). Group differences over time were analyzed using generalized estimating equations (GEEs) with all available data (i.e., Intent-To-Treat analyses). GEE results were followed-up with pairwise comparisons when applicable. Measures administered pre- and post-session (QSU and MNWS) were calculated as a change score and included as such in GEE analyses. Pre-session scores were subtracted from post session scores such that negative scores reflect decreases in withdrawal symptoms or smoking urges throughout the session. For measures administered at two or less time points, *t*-tests were used to examine group differences.